CLINICAL TRIAL: NCT06254274
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2 Study Evaluating the Safety, Tolerability, and Efficacy of RAY1225 in Participants With Type 2 Diabetes
Brief Title: A Study of RAY1225 in Participants With Type 2 Diabetes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAY1225-23-03
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RAY1225 (cohort 1) (Experimental): Participants received dose1 or dose2 RAY1225 administered subcutaneously (SC) once two week for 24 weeks.
  Interventions: Drug: RAY1225
- Placebo (cohort 1) (Placebo Comparator): Participants received Placebo administered SC once two weeks for 24 weeks.
  Interventions: Drug: Placebo
- RAY1225 (cohort 2) (Experimental): Escalating doses of RAY1225 administered subcutaneously (SC) once two week
  Interventions: Drug: RAY1225
- Placebo (cohort 2) (Placebo Comparator): Participants received Placebo administered SC once two week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAY1225 — Administered SC
  Arms: RAY1225 (cohort 1); RAY1225 (cohort 2)
Drug: Placebo — Administered SC
  Arms: Placebo (cohort 1); Placebo (cohort 2)

SUMMARY:
The main purpose of this study is to learn more about the Tolerability of RAY1225 in participants with type 2 diabetes mellitus. The study will also explore the efficacy of RAY1225. The study will last about six months for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes had been diagnosed for at least 12 weeks prior to screening and one of the following conditions:

   1. have T2DM controlled with diet and exercise alone;
   2. are stable in dose and type on a single or in a combination of oral antidiabetic medication, metformin, α-glucosidase inhibitors or SGLT-2 inhibitors only ,within 12 weeks before screening;
2. BMI ≥ 20 kg/m²；
3. Fasting blood-glucose（FPG）<15 mmol/L;
4. Weight change < 5% in the 12 weeks before screening;
5. Participants (including partners) must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product.

Exclusion Criteria:

1. have type 1 diabetes mellitus；
2. Severe diabetic complications, including proliferative retinopathy or maculopathy, severe diabetic neuropathy (e.g., urinary retention, urinary incontinence, and painful peripheral neuropathy), resting tachycardia, orthostatic hypotension, intermittent claudication, or diabetic foot;
3. Two or more episodes of ketoacidosis, lactic acidosis, or hyperosmolar state leading to hospitalization within 24 weeks before screening;
4. had grade 3 hypoglycemic events within 12 months before screening,
5. Three or more grade 2 hypoglycemic events occurred within 3 months before screening;
6. Have symptoms related to hypoglycemia at screening;
7. Within 6 weeks before screening, serious trauma, serious infection, or surgery that may have affected glycemic control was reported;
8. Have a family or personal history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia (MEN) Syndrome type 2 or with thyroid nodules of unknown etiology found at screening and considered clinically significant by the investigator.
9. Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty if performed >1 year prior to screening)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) | Baseline,Week 26
  HbA1c is the glycosylated fraction of hemoglobin A.

SECONDARY OUTCOMES:
Percentage of Participants With HbA1c Target Value of <6.5% | Baseline,Week26
Percentage of Participants With HbA1c Target Value of <7% | Baseline,Week26
Percentage of Participants With HbA1c Target Value of <5.7% | Baseline,Week26
Change From Baseline in Fasting Serum Glucose | Baseline,Week26

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijingcun, Hebei, China